CLINICAL TRIAL: NCT05404529
Title: A Phase 1 Open-label Trial to Evaluate the Pharmacokinetics and Safety Following Single Dose of Tavapadon in Participants With Mild and Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Brief Title: To Evaluate the Pharmacokinetics (PK) and Safety of Tavapadon in Participants With Mild and Moderate Hepatic Impairment Compared to Participants With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVL-751-1003
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Hepatic Impairment
Keywords: Healthy Volunteer; Mild Hepatic Impairment; Moderate Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate Hepatic Function (Experimental): Participants will receive a single dose of tavapadon, 0.5 milligrams (mg) or 0.25 mg tablet based on tolerability, on Day 1.
  Interventions: Drug: Tavapadon
- Mild Hepatic Function (Experimental): Participants will receive a single dose of tavapadon, 0.5 mg or 0.25 mg tablet based on tolerability, on Day 1.
  Interventions: Drug: Tavapadon
- Normal Hepatic Function (Experimental): Participants will receive a single dose of tavapadon, 0.5 mg or 0.25 mg tablet based on tolerability, on Day 1.
  Interventions: Drug: Tavapadon

INTERVENTIONS:
Drug: Tavapadon — Oral tablets
  Other Names: CVL-751

SUMMARY:
The primary purpose of the study is to assess the effect of hepatic impairment on the PK of tavapadon following administration of a single oral dose in participants with mild and moderate hepatic impairment relative to age, body weight, and sex-matched participants with normal hepatic function.

ELIGIBILITY:
Key Inclusion Criteria:

1. Body mass index of ≥17.5 to 42.0 0 kilograms per meter square (kg/m^2), inclusive, and a total body weight >50 kilograms (kg) [110 pounds (lbs)].
2. Must meet the criteria for Class A or B of the modified Child-Pugh classification.
3. Stable hepatic disease defined as no clinically significant change in disease status in the last 28 days prior to the screening visit.
4. Previous alcohol abuse is permitted provided that the participant is willing and able to follow lifestyle guidelines and has a negative breath alcohol test at Screening and Check-in (Day -1).

Key Exclusion Criteria:

1. Receipt of severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) vaccine or booster within 7 days of planned dosing.
2. Have recently been diagnosed with symptomatic Coronavirus Disease 2019 (COVID-19) or test positive for COVID-19 within 30 days prior to signing the informed consent form (ICF).
3. Taking any prohibited medication prior to randomization or likely to require prohibited concomitant therapy.
4. Has received study drug in a clinical trial of Tavapadon within 12 months of signing the ICF.
5. Acute hepatitis.
6. Grade ≥2 hepatic encephalopathy.
7. Participants who have received an organ transplant or are currently waiting for an organ transplant and are listed on the national transplant list.
8. Primary biliary cholangitis or primary sclerosing cholangitis.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Tavapadon | pre-dose and at multiple timepoints post-dose up to Day 7
Area Under the Plasma Concentration-time Curve from Time Zero to t (AUC0-t) of Tavapadon | pre-dose and at multiple timepoints post-dose up to Day 7
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUCinf) of Tavapadon | pre-dose and at multiple timepoints post-dose up to Day 7

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and AEs by Severity | Day 1 up to Follow-up (Day 15)
Number of Participants with Clinically Significant Abnormalities in Electrocardiogram (ECG) Values | Day 1 up to Follow-up (Day 15)
Number of Participants with Clinically Significant Abnormalities in Vital Sign Values | Day 1 up to Follow-up (Day 15)
Number of Participants with Clinically Significant Abnormalities in Laboratory Values | Day 1 up to Follow-up (Day 15)
Number of Participants with Clinically Significant Abnormalities in Physical and Neurological Examination Results | Day 1 up to Follow-up (Day 15)
Number of Participants with Change in Columbia Suicide Severity Rating Scale (C-SSRS) Score | Day 1 up to Follow-up (Day 15)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Miami, Florida, Miami, Florida
  - Orlando, Florida, Orlando, Florida
  - San Antonio, Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No